CLINICAL TRIAL: NCT00004229
Title: A Phase I Surrogate Endpoint Trial of Human Recombinant Endostatin in Patients With Advanced Solid Tumors Amenable to Biopsy
Brief Title: Endostatin in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02314; MDA-ID-99201; NCI-T99-0087; CDR0000067471 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-01-28; First posted 2004-04-19 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2002-12

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — Endostatins

ARMS (1):
- Arm I (Experimental): Patients undergo a biopsy during prestudy and after the second course of treatment. Patients receive endostatin IV daily for 4 weeks. Patients on dose level 1-6 receive endostatin over 20 minutes. Patients on dose level 7 receive endostatin over 40 minutes, with no treatment on day 2 of the first course only. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of endostatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.
  Interventions: Biological: recombinant human endostatin

INTERVENTIONS:
Biological: recombinant human endostatin

SUMMARY:
Phase I trial to study the effectiveness of endostatin in treating patients who have advanced solid tumors. Endostatin may stop the growth of cancer by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the optimal biologic dose of endostatin in patients with advanced solid tumors.

II. Determine the safety and tolerability of this regimen in these patients. III. Determine the extent, frequency, and duration of tumor response in these patients on this regimen.

IV. Determine the pharmacokinetic profile and interpatient pharmacologic variability of this regimen in these patients.

V. Determine the recommended phase II dose and schedule of this regimen.

OUTLINE: This is a dose escalation study.

Patients undergo a biopsy during prestudy and after the second course of treatment. Patients receive endostatin IV daily for 4 weeks. Patients on dose level 1-6 receive endostatin over 20 minutes. Patients on dose level 7 receive endostatin over 40 minutes, with no treatment on day 2 of the first course only. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity. Cohorts of 3-6 patients receive escalating doses of endostatin until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

Patients are followed for 1 month.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven advanced solid tumor for which no standard curative therapy exists
* Must be amenable to biopsy At least 1 site of measurable disease outside of irradiated field
* No brain metastases by CT or MRI scan

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-1
* WBC greater than 3,000/mm3
* Absolute neutrophil count greater than 1,500/mm3
* Platelet count greater than 100,000/mm3
* Hemoglobin greater than 10 g/dL
* Bilirubin less than 1.5 times upper limit of normal (ULN)
* ALT and AST less than 2.0 times ULN
* PT/PTT less than 1.5 times ULN
* Creatinine less than 1.5 mg/dL OR creatinine clearance greater than 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No concurrent uncontrolled medical or psychiatric disorder
* No history of bleeding diathesis

PRIOR CONCURRENT THERAPY:

* No concurrent over the counter biologic agents (e.g., shark cartilage)
* At least 3 weeks since prior chemotherapy (6 weeks since nitrosoureas or mitomycin)
* No more than 3 prior chemotherapy regimens for metastatic or recurrent disease (ECOG 1)
* Prior adjuvant chemotherapy for nonmetastatic disease allowed
* Concurrent stable dose of hormone replacement therapy allowed
* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy
* At least 24 hours since minor surgery (e.g., central venous placement)
* At least 4 weeks since major surgery (e.g., laparotomy, thoracotomy, or craniotomy)
* At least 30 days since other prior investigational agents
* No concurrent herbal remedies
* No concurrent usage of products containing heparin
* No other concurrent anticancer therapy
* Concurrent multivitamins allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 1999-10; Primary Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy S. Herbst, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States